CLINICAL TRIAL: NCT05155267
Title: Biomonitoring of Internal Exposure to MNPLs (Micro and NanoPlastics), and Its Effects, in Blood of Patients With Chronic Kidney Disease (CKD)
Brief Title: Biomonitoring of Internal Exposure to MNPLs, and Its Effects, in Blood of Patients With Chronic Kidney Disease (CKD)
Status: Recruiting | Type: Observational
Sponsor: Ricard Marcos (Other)
Collaborators: Instituto Murciano de Investigación Biosanitaria Virgen de la Arrixaca (Other); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Sponsor-Investigator, Ricard Marcos, Professor, Universitat Autonoma de Barcelona
Organization: Universitat Autonoma de Barcelona (Other)
Other Study IDs: 1-1
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases; Microplastics; Nanoplastics; Genotoxic Damage
Keywords: CKD; MNPLs
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood, urine and feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Kidney disease participants (CKD)_HD: CKD submitted to hemodialysis (HD)
  Interventions: Other: Biomonitoring study to detect MNPLs in biological samples and study of their health effects
- Chronic Kidney disease participants (CKD)_PD: CKD non-submitted to hemodialysis (pre-dialysis:PD)
  Interventions: Other: Biomonitoring study to detect MNPLs in biological samples and study of their health effects
- Controls: Healthy participants
  Interventions: Other: Biomonitoring study to detect MNPLs in biological samples and study of their health effects

INTERVENTIONS:
Other: Biomonitoring study to detect MNPLs in biological samples and study of their health effects — Determination of MNPLs levels, genotoxic damage and immunological effects

SUMMARY:
Micro and nanoplastics (MNPLs) effects on human heath is still preliminary. Chronic kidney disease (CKD) participants, specially does patients submitted to hemodialysis, are a population high exposed to plastics. The objective of our research is to be able to detect MNPLs on biological fluids of hemodialysis patients as well as their potential genotoxic and immunological damage.

DETAILED DESCRIPTION:
The exponential increase in the production/use of plastic translates into a parallel increase of environmental plastic-waste that is continuously degraded into micro and nanoplastics (MNPLs). Information on the MNPLs' effects on human health is still preliminary and, furthermore, the limitations in current methodologies prevent accurate human exposure/risk assessment.

The study aims to analyse specific biomarkers of exposure to MNPLs in humans, as well as biomarkers of genetic damage, which will allow an association between exposure to these plastic materials and the optimisation of different techniques for the detection and characterisation of MNPLs.

The study will evaluate the effect of exposure to MNPLs, analysing the genotoxic damage, different biomarkers of exposure and the effects on microbiota, in different body samples (urine, blood and feces).

ELIGIBILITY:
Inclusion Criteria for Chronic Kidney Disease (CKD) submitted to Hemodialysis:

* Participant submitted to hemodialysis for more than 3 months
* Between 18 and 85 years old
* Stable haemoglobin (more than 10 gr/dl)
* Absence of infectious disease at the date of sample collection and for a period of more than two weeks
* Absence of active neoplasia
* Stable vascular access

Inclusion Criteria for Chronic Kidney Disease (CKD) pre-dialysis:

* No hemodialysis treatment
* Between 18 and 85 years old
* Stable haemoglobin (more than 10 gr/dl)
* Glomerular filtration ≤ 20 ml/min
* Absence of infectious disease at the date of sample collection and for a period of more than two weeks
* Absence of active neoplasia

Inclusion Criteria for controls :

* Between 18 and 85 years old (paired by gender, age and lifestyle to the CKD patients)
* Absence of chronic kidney disease or dialysis treatment
* Absence of chronic pathology (including neoplasia)
* Absence of infectious disease at the date of sample collection and for a period of more than two weeks
* Spanish residence

Exclusion Criteria for both groups of CKD patients:

* Clinical instability
* Life expectancy of less than 12 months
* Coagulation system disorders
* Participation in other clinical study
* Pregnancy
* Unsigned informed consent

Exclusion criteria for controls:

* Participation in other clinical study
* Pregnancy
* Unsigned informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project will study a minimum of 25 adult participants with chronic kidney disease, included and not included in an haemodialysis programme. A control group (at least 25 individuals), matched by gender, age and lifestyle with CKD participants will be also included.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Biomonitoring study to detect the presence of MNPLs in biological fluids | Up to 1 year
  Micro and nanoplastic and/or derivatives, would be evaluated. Characterization of possible biomarkers of early biological effects on human health
Study of the effects of MNPLs on immune system | Up to 1 year
  Impact evaluation of MNPLs on transcriptome, secretome and inflammatory signalling and inflammasome activation. Investigating the effect of MNPLs on the function of the immune system in vivo and in high-risk individuals
Genotoxicity effects of exposure to MNPLs | Up to 1 year
  Genotoxic, chromosome damage evaluation and oxidative DNA damage will be analysed by the Comet assay and the micronucleus assay

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Pelegrín, Principal Investigator — Instituto Murciano de Investigación Biosanitaria (IMIB); Juan Bernardo Cabezuelo, Study Chair — Hospital Clínico Universitario Virgen Arrixaca (Murcia); Laura Martínez, Study Chair — Hospital Clínico Universitario Virgen Arrixaca (Murcia)
Locations (1):
- Servicio Murciano de Salud, Murcia, Spain